CLINICAL TRIAL: NCT04218071
Title: Phase 2 Study of 9-ING-41, a Glycogen Synthase Kinase 3 Beta (GSK 3β) Inhibitor, as a Single Agent or Combined With Ruxolitinib, in Patients With Myelofibrosis
Brief Title: Actuate 1901: 9-ING-41 in Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1901
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Myelofibrosis
Keywords: primary myelofibrosis; post polycythemia vera myelofibrosis; post essential thrombocythemia myelofibrosis; Ruxolitinib; Jak2 inhibitors; glycogen synthase kinase 3 beta; GSK3beta; 9-ING-41
MeSH Terms: conditions — Primary Myelofibrosis; Hereditary Sensory and Autonomic Neuropathies | interventions — ruxolitinib; 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione

STUDY DESIGN:
Intervention Model Description: Patients will receive either single agent 9-ING-41 or 9-ING-41 plus Ruxolitinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 9-ING-41 (Experimental): 9-ING-41 is administered by intravenous infusion twice weekly at a dose of 9.3 mg/kg. Cycle duration is 28 days.
  Interventions: Drug: 9-ING-41
- 9-ING-41 plus Ruxolitinib (Experimental): 9-ING-41 9.3 mg/kg will be administered by intravenous infusion twice weekly for cycle durations of 28 days with Ruxolitinib at doses specified in the protocol as appropriate for patient's platelet count.
  Interventions: Drug: Ruxolitinib; Drug: 9-ING-41

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib at protocol-specified doses for given platelet count
  Other Names: Jakafi
  Arms: 9-ING-41 plus Ruxolitinib
Drug: 9-ING-41 — 9-
  Other Names: 9-ING-41 Compound

SUMMARY:
9-ING-41 has anti-cancer clinical activity while not causing myelosuppression, and has both pre-clinical anti-fibrotic activity and activity against myelofibrosis. This Phase 2 study will study its efficacy in patients with advanced myelofibrosis.

DETAILED DESCRIPTION:
9-ING-41 is a first-in-class, intravenously administered, maleimide-based, small molecule, potent selective GSK-3β inhibitor with significant pre-clinical and clinical anticancer activity. In the ongoing Actuate 1801 study in a cohort of over 90 patients with advanced refractory malignancies, 9-ING-41 has exhibited no significant toxicity, including no myelosuppression, and significant anti-tumor activity. 9-ING-41 also has significant pre-clinical ability to reverse pathologic fibrosis in multiple models of pulmonary and pleural fibrosis. Reversal of fibrosis by an anti-fibrotic agent in patients with advanced myelofibrosis (MF) has recently been demonstrated to be of clinical benefit. 9-ING-41 has the potential to act both as an anti-neoplastic agent (without causing myelosuppression) and an anti-fibrotic agent in patients with MF. The efficacy of Ruxolitinib is limited in many patients by the inability to tolerate adequate doses for an adequate duration with myelosuppression being a frequent dose limiting toxicity. 9-ING-41 may reduce the dose of Ruxolitinib needed for optimal therapeutic response and/or reverse myelosuppression so than an adequate dose of Ruxolitinib can be tolerated. Pre-clinical data show synergy in MF between 9-ING-41 and Ruxolitinib. This Phase 2 study is designed to evaluate the efficacy of 9-ING-41, as a single agent or in combination with Ruxolitinib, in patients with advanced, poor prognosis MF.

ELIGIBILITY:
Inclusion Criteria:

Patient -

1. Is able to understand and voluntarily sign a written informed consent and is willing and able to comply with the protocol requirements including scheduled visits, treatment plan, laboratory tests and other study procedures
2. Is aged ≥ 18 years
3. Has documented diagnosis of symptomatic primary MF, PPV-MF or PET-MF as defined by the World Health Organization classification
4. Is ineligible or unwilling to undergo stem cell transplantation at time of study entry
5. Has laboratory function within specified parameters per local laboratory (may be repeated):

   * Absolute neutrophil count (ANC) ≥ 100/mL; platelets ≥ 20,000/mL
   * Transaminases (AST/ALT) and alkaline phosphatase ≤ 3 (≤ 10 X the upper limit of normal (ULN) if considered to be MF-related) x ULN; bilirubin ≤ 1.5 x ULN (unless patient has Gilbert's Syndrome)
   * Serum amylase and lipase ≤ 1.5 x ULN
6. Has adequate performance status (PS): Eastern Co-operative Oncology Group (ECOG) PS 0-2
7. Has received the final dose of any of the following treatments/procedures with the specified minimum intervals before first dose of 9-ING-41 (unless in the opinion of the investigator and the study medical coordinator the treatments/procedures will not compromise patient safety or interfere with study conduct:

   * Chemotherapy, immunotherapy, or systemic radiation therapy - 14 days maximum, or ≥ 5 half-lives (whichever is shorter)
   * Surgery with general anesthesia - 7 days
8. Patients who are to receive 9-ING-41 plus Ruxolitinib must have attempted ≥12 weeks of Ruxolitinib therapy and required dose reductions/interruptions and/or had an inadequate response
9. Women of childbearing potential must have a negative baseline blood or urine pregnancy test within 72 hours of first study therapy. Women may be neither breastfeeding nor intending to become pregnant during study participation and must agree to use effective contraceptive methods (hormonal or barrier method of birth control, or true abstinence) for the duration of study participation and in the following 100 days after discontinuation of study treatment
10. Male patients with partners of childbearing potential must take appropriate precautions to avoid fathering a child from screening until 100 days after discontinuation of study treatment and use appropriate barrier contraception or true abstinence
11. Must not be receiving any other investigational product

Exclusion Criteria:

Patient -

1. Is pregnant or lactating
2. Is known to be hypersensitive to any of the components of 9-ING-41 or to the excipients used in its formulation
3. Has >10% blasts in peripheral blood or bone marrow biopsy
4. Has had a myocardial infarction within 12 weeks of the first dose of 9-ING-41
5. Has any medical and/or social condition which, in the opinion of the investigator or study medical coordinator would preclude study participation
6. Is considered to be a member of a vulnerable population (for example, prisoners)
7. Herbal preparations / medications are prohibited throughout the study. These herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), Gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and Ginseng. Patients should stop using cannabinoids or herbal preparations/medications at least 7 days prior to first dose of study treatment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Response rate | 3-24 months
  The percent of patients with response will be assessed at the protocol specified timepoints according to the Revised IWG-MRT and ELN Response Criteria for MF (2013)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Georgia Cancer Center, Augusta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - Weill Cornell Medicine | NewYork-Presbyterian Meyer Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Brown University, Providence, Rhode Island
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jeffers A, Qin W, Owens S, Koenig KB, Komatsu S, Giles FJ, Schmitt DM, Idell S, Tucker TA. Glycogen Synthase Kinase-3beta Inhibition with 9-ING-41 Attenuates the Progression of Pulmonary Fibrosis. Sci Rep. 2019 Dec 12;9(1):18925. doi: 10.1038/s41598-019-55176-w. PMID 31831767
- [Result] Kuroki H, Anraku T, Kazama A, Bilim V, Tasaki M, Schmitt D, Mazar AP, Giles FJ, Ugolkov A, Tomita Y. 9-ING-41, a small molecule inhibitor of GSK-3beta, potentiates the effects of anticancer therapeutics in bladder cancer. Sci Rep. 2019 Dec 27;9(1):19977. doi: 10.1038/s41598-019-56461-4. PMID 31882719
- [Result] Ding L, Madamsetty VS, Kiers S, Alekhina O, Ugolkov A, Dube J, Zhang Y, Zhang JS, Wang E, Dutta SK, Schmitt DM, Giles FJ, Kozikowski AP, Mazar AP, Mukhopadhyay D, Billadeau DD. Glycogen Synthase Kinase-3 Inhibition Sensitizes Pancreatic Cancer Cells to Chemotherapy by Abrogating the TopBP1/ATR-Mediated DNA Damage Response. Clin Cancer Res. 2019 Nov 1;25(21):6452-6462. doi: 10.1158/1078-0432.CCR-19-0799. Epub 2019 Sep 18. PMID 31533931
- [Result] Wu X, Stenson M, Abeykoon J, Nowakowski K, Zhang L, Lawson J, Wellik L, Li Y, Krull J, Wenzl K, Novak AJ, Ansell SM, Bishop GA, Billadeau DD, Peng KW, Giles F, Schmitt DM, Witzig TE. Targeting glycogen synthase kinase 3 for therapeutic benefit in lymphoma. Blood. 2019 Jul 25;134(4):363-373. doi: 10.1182/blood.2018874560. Epub 2019 May 17. PMID 31101621
- [Result] Ugolkov AV, Bondarenko GI, Dubrovskyi O, Berbegall AP, Navarro S, Noguera R, O'Halloran TV, Hendrix MJ, Giles FJ, Mazar AP. 9-ING-41, a small-molecule glycogen synthase kinase-3 inhibitor, is active in neuroblastoma. Anticancer Drugs. 2018 Sep;29(8):717-724. doi: 10.1097/CAD.0000000000000652. PMID 29846250
- [Result] Karmali R, Chukkapalli V, Gordon LI, Borgia JA, Ugolkov A, Mazar AP, Giles FJ. GSK-3beta inhibitor, 9-ING-41, reduces cell viability and halts proliferation of B-cell lymphoma cell lines as a single agent and in combination with novel agents. Oncotarget. 2017 Nov 11;8(70):114924-114934. doi: 10.18632/oncotarget.22414. eCollection 2017 Dec 29. PMID 29383130
- [Result] Ugolkov A, Qiang W, Bondarenko G, Procissi D, Gaisina I, James CD, Chandler J, Kozikowski A, Gunosewoyo H, O'Halloran T, Raizer J, Mazar AP. Combination Treatment with the GSK-3 Inhibitor 9-ING-41 and CCNU Cures Orthotopic Chemoresistant Glioblastoma in Patient-Derived Xenograft Models. Transl Oncol. 2017 Aug;10(4):669-678. doi: 10.1016/j.tranon.2017.06.003. Epub 2017 Jun 30. PMID 28672195
- [Result] Ugolkov A, Gaisina I, Zhang JS, Billadeau DD, White K, Kozikowski A, Jain S, Cristofanilli M, Giles F, O'Halloran T, Cryns VL, Mazar AP. GSK-3 inhibition overcomes chemoresistance in human breast cancer. Cancer Lett. 2016 Oct 1;380(2):384-392. doi: 10.1016/j.canlet.2016.07.006. Epub 2016 Jul 14. PMID 27424289
- [Result] Pal K, Cao Y, Gaisina IN, Bhattacharya S, Dutta SK, Wang E, Gunosewoyo H, Kozikowski AP, Billadeau DD, Mukhopadhyay D. Inhibition of GSK-3 induces differentiation and impaired glucose metabolism in renal cancer. Mol Cancer Ther. 2014 Feb;13(2):285-96. doi: 10.1158/1535-7163.MCT-13-0681. Epub 2013 Dec 10. PMID 24327518
- [Result] Boren J, Shryock G, Fergis A, Jeffers A, Owens S, Qin W, Koenig KB, Tsukasaki Y, Komatsu S, Ikebe M, Idell S, Tucker TA. Inhibition of Glycogen Synthase Kinase 3beta Blocks Mesomesenchymal Transition and Attenuates Streptococcus pneumonia-Mediated Pleural Injury in Mice. Am J Pathol. 2017 Nov;187(11):2461-2472. doi: 10.1016/j.ajpath.2017.07.007. PMID 29073967
- [Result] Anraku T, Kuroki H, Kazama A, Bilim V, Tasaki M, Schmitt D, Mazar A, Giles FJ, Ugolkov A, Tomita Y. Clinically relevant GSK-3beta inhibitor 9-ING-41 is active as a single agent and in combination with other antitumor therapies in human renal cancer. Int J Mol Med. 2020 Feb;45(2):315-323. doi: 10.3892/ijmm.2019.4427. Epub 2019 Dec 12. PMID 31894292